CLINICAL TRIAL: NCT02515812
Title: Comparative Study of Cardiac Adrenergic Function Explored by I-123-MIBG and CZT Camera (D-SPECT) Versus Anger Camera in Patients With Heart Failure
Acronym: ADRECARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-075
Record Dates: First submitted 2015-07-28; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Gamma Cameras

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adrenergic Function Explorations with CZT camera (Experimental): I-123-MIBG and CZT Camera (D-SPECT)
  Interventions: Drug: I-123-MIBG; Device: CZT Camera (D-SPECT)
- Adrenergic Function Explorations with Anger camera (Active Comparator): I-123-MIBG and Anger Camera
  Interventions: Drug: I-123-MIBG; Device: Anger Camera

INTERVENTIONS:
Drug: I-123-MIBG
Device: CZT Camera (D-SPECT)
  Arms: Adrenergic Function Explorations with CZT camera
Device: Anger Camera
  Arms: Adrenergic Function Explorations with Anger camera

SUMMARY:
Cardiological examination constitute one of the major directions in nuclear medicine for detection of myocardial ischemia in patients suspected of coronary disease. In Caen, they constitute 20% of the activity of nuclear medicine. Systolic heart failure (HF) ischemic or nonischemic origin represents a new area of activity of the nuclear cardiology. This is HF stratification study based on cardiac adrenergic function after injection of a tracer: I-123-MIBG. The team Caen nuclear cardiology is one of two teams recognized internationally in the field of evaluating the cardiac sympathetic innervation in cardiomyopathies. Numerous publications from 1992 to the present day have reported encouraging results for the daily use of this tracer in the evaluation of patients with LV dysfunction IC. Recently, interest in using the MIBG has been shown as a prognostic marker of HF in a prospective study of 961 patients. Typically, the camera used was an Anger camera with collimating Nai standard called parallel holes.

The main objective is to validate the measurements of cardiac adrenergic function evaluated by cardiopulmonary mediastinal reports and sympathetic innervation scores VG after injection of I-123-MIBG in 80 patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years (except major patients under guardianship)
* patient who signed the consent form
* written and spoken French
* Beneficiaries of the social security system
* Stable heart failure with LV dysfunction (<45%) of ischemic or nonischemic origin

Exclusion Criteria:

* Patients with a recent history (<21 days) acute coronary failure (myocardial infarction, unstable angina)
* Patients with severe extra-cardiac disease may interfere with treatment decisions (cancer, severe hepatic or renal impairment)
* Major patients under guardianship
* Pregnant or lactating women
* Women in age and condition of childbearing
* Patients unable to understand the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
SRSI (summed rest score innervation) | 4 hours after I-123-MIBG perfusion
  with CZT camera and Anger camera
SRS (summed rest score) | 4 hours after I-123-MIBG perfusion
  with CZT camera and Anger camera

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine Nucléaire -CHU de Caen, Caen, France